CLINICAL TRIAL: NCT06149715
Title: Evaluating Comparative Efficacy of Sawyer PointOne Filter Types in Ciudad Victoria, Mexico
Brief Title: Water Filter Study in Ciudad Victoria
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Aquora Research & Consulting, LLC (Industry)
Collaborators: Sawyer Products, Inc (Unknown); The Bucket Ministry (Unknown); Sparrow Data Solutions (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CiudadVictoriaFilterStudy
Record Dates: First submitted 2023-11-17; First posted 2023-11-29 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Waterborne Diseases; Diarrhea
MeSH Terms: conditions — Waterborne Diseases; Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bottle Filter Arm (Experimental): Receive a filter which attaches to a bottle. If the household does not have an eligible tap, they are randomly assigned to either this arm or the Bucket Filter Arm.
  Interventions: Device: Bottle Filter
- Bucket Filter Arm (Experimental): Receive a filter which attaches to a bucket. If the household does not have an eligible tap, they are randomly assigned to either this arm or the Bottle Filter Arm.
  Interventions: Device: Bucket Filter
- Tap Filter Arm (Experimental): All households with an eligible tap (compatible with filter and runs) will receive a tap filter.
  Interventions: Device: Tap Filter

INTERVENTIONS:
Device: Bottle Filter — The household is given a Sawyer Squeeze Water Filtration System.
  Arms: Bottle Filter Arm
Device: Bucket Filter — The household is given a Sawyer International Bucket System, which is a Squeeze Water Filtration System that is integrated with a hose and bucket.
  Arms: Bucket Filter Arm
Device: Tap Filter — The household is given a Sawyer Tap Water Filtration System.
  Arms: Tap Filter Arm

SUMMARY:
This study measures effects of water filters and filter types on household health in Ciudad Victoria, Mexico.

DETAILED DESCRIPTION:
A project to assess the water quality in Ciudad Victoria, Mexico and the effectiveness of different Sawyer PointOne Filter types (Bucket, Tap, Squeeze) . The project is designed to 1) assess the impact of filters on health and well-being of families, 2) assess the impact of filters on the economic status of families and 3) compare different filter formats for use/adoption on the above metrics. The project will provide information about how well the different filters are working in urban households in a middle-income Latin American country, make recommendations for future deployment of filter types in similar settings, and determine the potential for scaling the use of filter systems to provide clean drinking water for people in need in future projects.

ELIGIBILITY:
Inclusion Criteria:

* Recruiting will occur in Ciudad Victoria, Mexico at any household in the areas surveyed

Exclusion Criteria:

* None, except those who decline the survey and/or filter

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported diarrhea rates from initial filter distribution to end of follow up | 3 months follow up
  Self-reported diarrhea rates in households surveyed at distribution of the water filter and at each follow up visit.

SECONDARY OUTCOMES:
Change in other self-reported health outcomes from distribution to end of follow up | 3 months follow up
  Other health outcomes related to waterborne illness (such as fever, vomiting, muscle aches, rashes, etc.) which are also self-reported in the household surveys.
Change in household economic outcomes from distribution to end of follow up | 3 months of follow up
  Household economic outcomes related to costs of water and waterborne illnesses (such as money spent on water, money spent on medical costs, days of work missed due to diarrhea, etc.) which are also self-reported in the household surveys.

CONTACTS AND LOCATIONS:
Locations (1):
- Ciudad Victoria, Ciudad Victoria, Mexico

IPD SHARING:
Plan to Share IPD: No